CLINICAL TRIAL: NCT05476159
Title: Anastomotic Leak Test Using Indocyanine Green During Laparoscopic Roux-en-y Gastric Bypass
Brief Title: Indocyanine Green Test in Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Medical doctor, University of Foggia
Other Study IDs: 5
Record Dates: First submitted 2022-07-23; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Obesity, Morbid; Surgery; Leak, Anastomotic
MeSH Terms: conditions — Obesity, Morbid; Anastomotic Leak | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Drug: Indocyanine green solution — Adequate perfusion was defined as "the direct and clear visualization of the fluorescence along the gastric tube, relative to the excised specimen, after an estimated time of 150-180 s after i.v. administration injection
Device: Gastric bypass — Roux and Y Gastric bypass

SUMMARY:
Indocyanine green (ICG) can be injected into the human bloodstream and it allows us to show stomach vascularity in real time

ELIGIBILITY:
Inclusion Criteria:

* BMI>40kg/m2

Exclusion Criteria:

* Non obese patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The aim of our study is to observe the preliminary results of the application of indocyanine green fluorescence (IGF) during laparoscopic Roux-en-Y Gastric Bypass (RYGB in our center and how the perfusion of the gastro-jejunal anastomosis affects the onset of fistula.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Positive Intraoperative Indocyanine green test | During surgery (within 150-180 minutes)
  Intraoperative indocyanine green test was performed

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Pavone, Principal Investigator — University of Foggia
Locations (1):
- University of Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavone G, Fersini A, Pacilli M, Cianci P, Ambrosi A, Tartaglia N. Anastomotic leak test using indocyanine green during laparoscopic Roux-en-Y gastric bypass: A cohort study. Ann Med Surg (Lond). 2022 Nov 17;84:104939. doi: 10.1016/j.amsu.2022.104939. eCollection 2022 Dec. PMID 36536736

DOCUMENTS (1):
  • Study Protocol (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT05476159/Prot_000.pdf